CLINICAL TRIAL: NCT03585374
Title: Efficacy and Safety of Methoxyflurane Vaporized (PENTHROX®) in the Treatment of Acute Trauma Pain in Pre-hospital Setting and in the Emergency Department in Italy: a Multicentre, Randomized, Controlled, Open-label Study
Brief Title: Trauma Acute Pain Treatment With Methoxyflurane Vaporized (PENTHROX®): Efficacy and Safety Study (MEDITA)
Acronym: MEDITA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Pharmaceuticals srl (Industry)
Collaborators: Bioikos Ambiente Srl (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR311-3504
Record Dates: First submitted 2018-05-31; First posted 2018-07-13 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2018-12

CONDITIONS: Acute Traumatic Pain
Keywords: pain; methoxyflurane; Penthrox
MeSH Terms: conditions — Pain | interventions — Methoxyflurane; Morphine; Acetaminophen; Ketoprofen

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned to Penthrox (test group) or standard analgesic treatment (comparison group). As per local clinical practice, the standard analgesic will vary according to pain intensity score measured by Numerical Rating Scale (NRS): morphine, in case of score ≥ 7 or paracetamol/ketoprofen in case of score 4-6. Penthrox treatment will be performed by inhalatory route and will last maximum 25 minutes. the standard of care will be administered by an intravenous drip lasting at maximum 10 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A_test drug_Methoxyflurane (Penthrox®) (Experimental): Pain from moderate to severe (NRS score 4-10). 3 ml of methoxyflurane vaporized through the Penthrox® inhaler. The drug is self administered under the supervision of investigators/study nurse. The treatment duration is about 25 minutes. The patient is instructed to breath normally and to close the diluter aperture via his/her forefinger to increase the analgesic effect, if needed. In case of pain increase or insufficient pain relief the investigator is allowed to administer a rescue medication as per local routine practice.
  Interventions: Combination Product: Methoxyflurane and Penthrox inhaler
- B_comparator_Morphine/Paracetamol/Ketoprofen (Active Comparator): The comparator to be administered will vary according to pain intensity and local clinical practice.
  In case of severe pain (NRS score ≥ 7), morphine will be administered at a dose of 0.10 mg/kg body weight.
  In case of moderate pain (NRS score 4-6) paracetamol or ketoprofen will be administered respectively at a 1 g and 100 mg dose.
  All comparator will be administered by intravenous drip in a maximum 10 minutes time of infusion. .
  Maximum time of infusion 10 minutes.
  Interventions: Drug: Morphine; Drug: Paracetamol; Drug: Ketoprofen

INTERVENTIONS:
Combination Product: Methoxyflurane and Penthrox inhaler — 3ml of methoxyflurane vaporized through an inhaler (Penthrox). Inhalation, by regular breathing, last about 25 minutes.
  Other Names: Penthrox
  Arms: A_test drug_Methoxyflurane (Penthrox®)
Drug: Morphine — Each site will use the commercial available product already in use as per local clinical practice. The drug will be intravenously administered at a dose of 0.10 mg/Kg body weight. The time of infusion should be not longer than 10 minutes.
  Other Names: Morphine for intravenous use
  Arms: B_comparator_Morphine/Paracetamol/Ketoprofen
Drug: Paracetamol — Each site will use the commercial available product already in use as per local clinical practice. The drug will be intravenously administered at a 1 g dose The time of infusion should be not longer than 10 minutes.
  Other Names: Paracetamol for intravenous use
  Arms: B_comparator_Morphine/Paracetamol/Ketoprofen
Drug: Ketoprofen — Each site will use the commercial available product already in use as per local clinical practice. The drug will be intravenously administered at a 100 mg dose. The time of infusion should be not longer than 10 minutes.
  Other Names: Ketoprofen for intravenous use
  Arms: B_comparator_Morphine/Paracetamol/Ketoprofen

SUMMARY:
The prompt treatment of pain due to minor trauma is often an unmet need in both Emergency Room Department and Ambulance Rescue. Most of the available drugs are intravenously administered and such route of administration may account for delay in the pain relief onset.

Methoxyflurane is an halogenated anesthetic, self-administered by the patient at sub-anesthetic dose through an easy to handle inhaler (Penthrox®). The efficacy and safety of Penthrox® in the treatment of acute traumatic pain will be investigated in an out-of-hospital and in hospital emergency medical care setting.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be provided by each patient prior to any study-specific activity. In cases where the patient is unable to write autonomously, it must be obtained a verbal consent in presence of a witness that the patient will have to confirm autonomously as soon as (s)he is able
* Stable, vigilant and collaborative patient i.e. able to understand and communicate with the examiner in order to carry out the study activities
* Age ≥ 18 years
* Trauma to the limbs (fracture, dislocation, crushing, bruising) in a single district.

N.B. For recruiting, given the particular setting, no instrumental confirmation is required but suspicion of involvement of a single district is sufficient.

- Moderate to severe pain, detected by the Numerical Rating Scale (NRS score ≥4)

Exclusion Criteria:

* Personal or family history (parents or siblings) for malignant hyperthermia.
* History of severe adverse reactions to inhaled anesthetics.
* History of renal failure
* History of liver failure.
* Trauma risky dynamics (ejection from the vehicle, cabin deformation, death of an occupant of the same vehicle, motor vehicle / pedestrian or cyclist impact with a motor vehicle in motion, projection / overturn, fall from a height of> 3 meters, extraction on event place > 20 min).
* Altered level of vigilance and / or conscience (GCS <15)
* Symptomatic hypotension or Systolic Pressure <100 mm / Hg
* Discomfort with Respiratory Rate > 20 and Oxygen Saturation <95%
* Known pregnancy status.Note: a 1 day delay with respect to the planned menstruation date (28days since the beginning of the previous one) has to be considered a suspected pregnancy.
* Hypersensitivity to methoxyflurane, to any fluorinated anesthetic or to the E321 butylhydroxytoluene excipient.
* Current treatment with any analgesic for chronic pain or in the previous 5 hours (8 hours in the case of diclofenac).
* Known allergy to both paracetamol and non-steroidal anti-inflammatory drugs or known hypersensitivity to morphine
* All types of acute abdomen and paralytic ileus
* Hearth failure
* Recent (within2 months) biliary tract surgery
* Current bronchial asthma attack
* Uncontrolled epilepsy
* Depressive state treated with Monoamine Oxidase Inhibitors (ongoing or interrupted less 3 wks ago)
* Treatment with naltrexone
* History of active or recurrent peptic ulcer/hemorrhage (2 or more episodes of documented ulceration or bleeding in the last 6 months)
* Bleeding diathesis
* Current Intensive diuretic therapy
* Chronic dyspepsia, gastritis with significant episodes in the last 2 months
* Leucopenia and thrombocytopenia, current hemorrhages
* Current anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Change in the intensity of pain within 10 minutes. | From baseline up to 10 minutes later.
  The change in the pain intensity occurring from baseline (patient randomization) up to 10 minutes later. The pain intensity is measured by a 100 mm Visual-Analogic Scale (VAS). The pain intensity is measured at the baseline and after 3, 5, 10 minutes and the difference with the baseline measure is calculated. The changes (differences) from baseline will be compared between the two arms regardless the class of intensity pain (moderate + severe) and for the class of moderate pain.

SECONDARY OUTCOMES:
Need for rescue medication. | From baseline up to 30 minutes later.
  Percentage of patients who are using rescue medication for insufficient or unsatisfactory therapeutic effect of the trial drugs.
Change in the intensity of pain within 30 minutes. | From baseline up to 30 minutes later.
  The change in the pain intensity occurring from baseline up to 30 minutes later. The pain intensity is measured by a 100 mm Visual-Analogic Scale (VAS). The pain intensity is measured after 15, 20, 25, 30 minutes from baseline and the difference with the baseline measure is calculated. The changes (differences) from baseline will be compared between the two arms regardless the class of intensity pain (moderate + severe).
Time to pain relief. | From baseline up to 30 minutes.
  Time to get relief from pain starting from randomization. The patient will be asked to refer when he/she feel better.
Global assessment of treatment efficacy perceived by the patient. | From baseline to 30 minutes later or to the end of the treatment (whichever occurs first).
  30 minutes after randomization the patient will be asked to rate according to a 5 levels Likert scale (poor, moderate, good, very good, excellent) the global efficacy of the treatment.
Global assessment of treatment practicality in the investigator's opinion. | From baseline to 30 minutes later or to the end of the treatment (whichever occurs first).
  30 minutes after randomization the treating investigator will be asked to rate according to a 5 levels Likert scale (poor, moderate, good, very good, excellent) the practicality of the administered treatment.
Need for dilution hole closure (only Experimental Arm). | From baseline up to 30 minutes later.
  The closure of the dilution hole of the Penthrox device increases the inhalated amount of methoxyflurane and its antalgic effect. The patient will be instructed about the chance to close that hole and will be asked to refer the occurrence.
Change in the intensity of pain within 30 minutes by trauma type. | From baseline up to 30 minutes later.
  The change in the pain intensity occurring from baseline (patient randomization) up to 30 minutes later. The pain intensity is measured by a 100 mm Visual-Analogic Scale (VAS). The pain intensity is measured at the baseline and after 3, 5, 10, 15, 20, 25, 30 minutes and the difference with the baseline measure is calculated. The changes (differences) from baseline to each of the following timepoints for each trauma type will be compared between the two arms regardless the class of intensity pain (moderate + severe).
Incidence of Treatment-Emergent Adverse Events (AE) | From baseline up to 16 days later.
  Each untoward clinical event not related, in the Investigator judgement, to the underlying patient inclusion condition (trauma) will be recorded. Seriousness, relationship with the investigational drug, action taken for AE treatment will recorded for each AE.
Change in pulse rate | From baseline up to 30 minutes later.
  The pulse rate (beats/min) will be measured (either manually or automatically) at baseline and 10, 30 minutes later. The difference between the baseline values and the following ones will be calculated.
Change in blood pressure | From baseline up to 30 minutes later.
  The Blood Systolic and Diastolic pressure (mmHg) will be measured at baseline and 10, 30 minutes later. The difference between the baseline values and the following ones will be calculated.
Change in respiration rate | From baseline up to 30 minutes later.
  The respiration rate (breaths/min) will be measured (either manually or automatically) at baseline and 10, 30 minutes later. The difference between the baseline values and the following ones will be calculated.
Incidence of treatment-emergent pregnancy | From baseline up to 16 days later. The follow-up until delivery is out from the scope of the trial.
  Pregnant patients or suspected to be pregnant are excluded from the trial. In case of occurrence the pregnancy will be recorded and followed up until delivery for pharmacovigilance purposes.
Incidence of investigational medicinal drug misuse/abuse | From baseline up to 30 minutes later or to the end of the treatment (whichever occurs first).
  The occurrence of Investigational medicinal drug abuse (persistent or sporadic, intentional excessive use of medicinal products which is accompanied by harmful physical or psychological effects) or misuse (intentionally and inappropriately use not in accordance with the prescribed dose) during the treatment phase will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Germana Ruggiano, Dr, Principal Investigator — Azienda Sanitaria di Firenze Ospedale Santa Maria Annunziata DEA -Medicina D'Urgenza
Locations (16):
- Italy (16):
  - AO Universitaria- Policlinico V.Emanuele Medicina e Chirurgia d'Accettazione e d'Urgenza, Catania, CT
  - AO per l'Emergenza- Cannizzaro UO Servizio di Urgenza Emergenza Sanitaria 118, Catania, CT
  - Medicina D'Urgenza ed Accettazione Azienda Ospedaliera di Catanzaro "Pugliese-Ciaccio", Catanzaro, CZ
  - Azienda USL della Romagna - Forlì Unità Operativa Pronto Soccorso, Medicina d'Urgenza, 118, Forlì, FC
  - Azienda Sanitaria di Firenze Ospedale Santa Maria Annunziata DEA -Medicina D'Urgenza, Bagno a Ripoli, FI
  - AUSL della ROMAGNA Ospedale M. Bufalini Pronto Soccorso - Medicina d'Urgenza, Cesena, Forlì-Cesena
  - IRCCS San Martino Servizio 118, Genova, GE
  - Istituto Clinico Humanitas - Pneumologia e Medicina d'urgenza, Rozzano, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico Dipartimento di Anestesia e Terapia Intensiva Donna-Bambino, Milan, MI
  - ULSS 6 EUGANEA ex Ulss 16 Pronto Soccorso e Medicina d'Urgenza Ospedale S. Antonio, Padua, PD
  - OSPEDALE DI FAENZA Pronto Soccorso - Medicina d'Urgenza, Faenza, Ravenna
  - AOU (Azienda Ospedaliera Universitaria) Sassari Unità Operativa Complessa Medicina d'Accettazione e d'Urgenza - P.S. - O.B.I., Sassari, SS
  - ATS (Azienda tutela Salute)_Struttura Complessa Centrale Operativa 118, Sassari, SS
  - Medicina e Chirurgia di accettazione e di urgenza Humanitas Gradenigo - Presidio Sanitario, Torino, TO
  - Azienda USL Toscana Centro U.O. Centrale Operativa 118, Pistoia
  - AUSL della ROMAGNA Ospedale degli Infermi U.O. Pronto Soccorso - Medicina d'Urgenza, Rimini

REFERENCES:
- [Background] Todd KH, Ducharme J, Choiniere M, Crandall CS, Fosnocht DE, Homel P, Tanabe P; PEMI Study Group. Pain in the emergency department: results of the pain and emergency medicine initiative (PEMI) multicenter study. J Pain. 2007 Jun;8(6):460-6. doi: 10.1016/j.jpain.2006.12.005. Epub 2007 Feb 15. PMID 17306626
- [Background] Guru V, Dubinsky I. The patient vs. caregiver perception of acute pain in the emergency department. J Emerg Med. 2000 Jan;18(1):7-12. doi: 10.1016/s0736-4679(99)00153-5. PMID 10645828
- [Background] Brown JC, Klein EJ, Lewis CW, Johnston BD, Cummings P. Emergency department analgesia for fracture pain. Ann Emerg Med. 2003 Aug;42(2):197-205. doi: 10.1067/mem.2003.275. PMID 12883507
- [Background] Rupp T, Delaney KA. Inadequate analgesia in emergency medicine. Ann Emerg Med. 2004 Apr;43(4):494-503. doi: 10.1016/j.annemergmed.2003.11.019. PMID 15039693
- [Background] Berben SA, Schoonhoven L, Meijs TH, van Vugt AB, van Grunsven PM. Prevalence and relief of pain in trauma patients in emergency medical services. Clin J Pain. 2011 Sep;27(7):587-92. doi: 10.1097/AJP.0b013e3182169036. PMID 21505324
- [Background] Dale J, Bjornsen LP. Assessment of pain in a Norwegian Emergency Department. Scand J Trauma Resusc Emerg Med. 2015 Oct 29;23:86. doi: 10.1186/s13049-015-0166-3. PMID 26514633
- [Background] Mills AM, Shofer FS, Chen EH, Hollander JE, Pines JM. The association between emergency department crowding and analgesia administration in acute abdominal pain patients. Acad Emerg Med. 2009 Jul;16(7):603-8. doi: 10.1111/j.1553-2712.2009.00441.x. Epub 2009 Jun 22. PMID 19549018
- [Background] Pines JM, Hollander JE. Emergency department crowding is associated with poor care for patients with severe pain. Ann Emerg Med. 2008 Jan;51(1):1-5. doi: 10.1016/j.annemergmed.2007.07.008. Epub 2007 Oct 25. PMID 17913299
- [Background] Dayan AD. Analgesic use of inhaled methoxyflurane: Evaluation of its potential nephrotoxicity. Hum Exp Toxicol. 2016 Jan;35(1):91-100. doi: 10.1177/0960327115578743. Epub 2015 Apr 28. PMID 25926525
- [Background] Tomi K, Mashimo T, Tashiro C, Yagi M, Pak M, Nishimura S, Nishimura M, Yoshiya I. Alterations in pain threshold and psychomotor response associated with subanaesthetic concentrations of inhalation anaesthetics in humans. Br J Anaesth. 1993 Jun;70(6):684-6. doi: 10.1093/bja/70.6.684. PMID 8329263
- [Background] Coffey F, Wright J, Hartshorn S, Hunt P, Locker T, Mirza K, Dissmann P. STOP!: a randomised, double-blind, placebo-controlled study of the efficacy and safety of methoxyflurane for the treatment of acute pain. Emerg Med J. 2014 Aug;31(8):613-8. doi: 10.1136/emermed-2013-202909. Epub 2014 Apr 17. PMID 24743584
- [Background] Grindlay J, Babl FE. Review article: Efficacy and safety of methoxyflurane analgesia in the emergency department and prehospital setting. Emerg Med Australas. 2009 Feb;21(1):4-11. doi: 10.1111/j.1742-6723.2009.01153.x. PMID 19254307
- [Background] Jacobs IG. Health effects of patients given methoxyflurane in the prehospital setting: a data linkage study. The Open Emergency Medicine Journal 3: 7-13, 2010.
- [Derived] Serra S, Voza A, Ruggiano G, Fabbri A, Bonafede E, Sblendido A, Soldi A, Farina A; MEDITA Study Group. Efficacy, Practicality, and Safety of Inhaled Methoxyflurane in Elderly Patients with Acute Trauma Pain: Subgroup Analysis of a Randomized, Controlled, Multicenter, Open-Label Trial (MEDITA). J Pain Res. 2020 Jul 16;13:1777-1784. doi: 10.2147/JPR.S255532. eCollection 2020. PMID 32765053
- [Derived] Mercadante S, Voza A, Serra S, Ruggiano G, Carpinteri G, Gangitano G, Intelligente F, Bonafede E, Sblendido A, Farina A, Soldi A, Fabbri A; MEDITA Study Group. Analgesic Efficacy, Practicality and Safety of Inhaled Methoxyflurane Versus Standard Analgesic Treatment for Acute Trauma Pain in the Emergency Setting: A Randomised, Open-Label, Active-Controlled, Multicentre Trial in Italy (MEDITA). Adv Ther. 2019 Nov;36(11):3030-3046. doi: 10.1007/s12325-019-01055-9. Epub 2019 Oct 12. PMID 31612359
- [Derived] Fabbri A, Carpinteri G, Ruggiano G, Bonafede E, Sblendido A, Farina A, Soldi A; MEDITA Study Group. Methoxyflurane Versus Standard of Care for Acute Trauma-Related Pain in the Emergency Setting: Protocol for a Randomised, Controlled Study in Italy (MEDITA). Adv Ther. 2019 Jan;36(1):244-256. doi: 10.1007/s12325-018-0830-x. Epub 2018 Nov 22. PMID 30467809
- See also: Penthrox Summary of Product Characteristics — https://www.medicines.org.uk/emc/product/1939/smpc